CLINICAL TRIAL: NCT06211790
Title: Proteomic Guided First-line Precision Treatment of Renal Clear Cell Carcinoma: a Single-center, Prospective, Phase II Umbrella Clinical Study
Brief Title: Proteomic Guided First-line Precision Treatment of Renal Clear Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Upcoming
Record Dates: First submitted 2024-01-03; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma; Renal Clear Cell Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — anlotinib; Everolimus; tislelizumab

STUDY DESIGN:
Intervention Model Description: patients with renal cell carcinoma will be divided into three types, FuDan-GP1 subtype (targeted sensitive type), FuDan-GP2 subtype (Cold tumor) and FuDan-GP3 subtype (progenitor infiltrating type) in accordance with the condition of response to TKIs and the infiltration of immune cells, which dates from previous protein genomics study published by Nature Communications.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FuDan-GP1 subtype (Experimental): FuDan-GP1 subtype is targeted sensitive type. Treatment regimen：anlotinib 12 mg PO, QD, 14 days on - 7 days off.
  Interventions: Drug: Anlotinib, Everolimus and Tislelizumab
- FuDan-GP2 subtype (Experimental): FuDan-GP2 subtype is Cold tumor type. Treatment regimen：anlotinib 12 mg PO, QD, 14 days on - 7 days off combined with everolimus 5 mg PO, QD.
  Interventions: Drug: Anlotinib, Everolimus and Tislelizumab
- FuDan-GP3 subtype (Experimental): FuDan-GP3 subtype is progenitor infiltrating type. Treatment regimen：anlotinib 12 mg PO, QD, 14 days on - 7 days off combined with tislelizumab 200 mg, IV, Q3W.
  Interventions: Drug: Anlotinib, Everolimus and Tislelizumab

INTERVENTIONS:
Drug: Anlotinib, Everolimus and Tislelizumab — Anlotinib (PO, QD), Everolimus (PO, QD) and Tislelizumab (IV, Q3W)

SUMMARY:
Based on different subtypes, subjects will be placed in one of three treatment groups to explore individual efficacy and safety of various treatment regimen.

DETAILED DESCRIPTION:
MSKCC Prognostic Model and IMDC(International Metastatic Renal Cell Carcinoma Database Consortium) Criteria are derived from cytokine and targeted therapy era, separately. In order to adapt to immunotherapy era and achieve the precision treatment in patients with kidney cancer, a new molecular typing map is urgent to be set up. In this study, patients with renal cell carcinoma will be divided into three types, FuDan-GP1(glycoprotein I) subtype (targeted sensitive type), FuDan-GP2(glycoprotein 2) subtype (Cold tumor) and FuDan-GP3(glycoprotein 3) subtype (progenitor infiltrating type) in accordance with the condition of response to TKIs(tyrosine kinase inhibitor) and the infiltration of immune cells, which dates from previous protein genomics study published by Nature Communications. Based on the gene proteomic analysis of tissue samples, a molecular typing map was set up and the efficacy and safety of anlotinib, anlotinib combined with everolimus, and anlotinib combined with tislelizumab in the first-line treatment of unresectable or metastatic renal clear cell carcinoma will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria are eligible to participate in the trial:

* Male or female aged 18 and ≤ 75;
* Histologically or cytologically confirmed unresectable or metastatic clear cell carcinoma of the kidney, which may contain sarcomatoid lesions;
* At least one measurable target lesion at the time of enrollment according to RECIST1.1(Response Evaluation Criteria In Solid Tumors) standards;
* Tissue samples are available for testing;
* No previous systemic treatment for the disease;
* ECOG(Eastern Cooperative Oncology Group) PS(performance status) 0-1;
* Normal function of major organs (14 days prior to enrollment), i.e. meeting the following criteria:

  1. Blood routine examination criteria should be met (no blood transfusion and no granulocyte colony were received within 14 days before enrollment Stimulator therapy) :

     HB 90 g/L or higher The ANC(absolute neutrophil count) acuity 1.5 x 109 / L PLT(platelet count) acuity 100 x 109 / L
  2. No functional organic disease, the following criteria should be met:

Serum creatinine (Cr) ≤ 1.5× upper limit of normal (ULN) or creatinine clearance ≥40 mL/min T-bil ≤1.5×ULN upper limit of normal value ALT(Alanine transaminase) and AST≤2.5×ULN If liver metastasis, ALT and AST≤5×ULN

* Expected survival ≥3 months;
* Patients with potential fertility need to use contraception during the study period;
* Patients who volunteered to participate in this study and signed informed consent.

Exclusion Criteria:

Patients with any of the following conditions will be excluded from the trial:

1. Patients who have received the following medical interventions in the four weeks prior to treatment:

   * Radiation, surgery, chemotherapy, immunotherapy or molecular targeted therapy for tumors
   * To participate in other clinical studies of drug therapy
   * Live attenuated vaccine history
2. Previously received PD-1/PD-L1 monoclonal antibody, CTLA-4 antibody(cytolytic T lymphocyte-associated antigen) or other immunotherapy;
3. Previously received targeted therapy;
4. Definite brain/meningeal metastasis;
5. Patients who received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive drugs within 14 days prior to enrollment;
6. Any active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism), or known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
7. Severe disturbances (CTCAE, Common Terminology Criteria for Adverse Events> Class 2) occurred within 4 weeks prior to administration of the study drug;Baseline chest imaging suggests active pulmonary inflammation, signs and symptoms of infection (unexplained fever >38.5 degrees) within 14 days prior to first use of the study drug, or the need for oral or intravenous antibiotic treatment;
8. Patients with clinically significant bleeding symptoms or definite bleeding tendency within 3 months prior to treatment, or with arteriovenous thrombosis events occurring within 6 months prior to treatment;
9. Active cardiovascular disease, such as myocardial infarction, severe/unstable angina, or New York Heart Association Class III or IV congestive heart failure, was present in the 6 months prior to treatment.
10. Have had other malignancies in the past 5 years (basal cell carcinoma of the skin that has been cured, except carcinoma in situ of the breast and carcinoma in situ of the cervix);
11. Have multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
12. Known to have active tuberculosis;
13. HIV antibody positive, active hepatitis B or C (HBV, HCV);
14. Is known to be allergic to the investigational drug or any excipients thereof, or has had a severe allergic reaction to other monoclonal antibodies;
15. Pregnant or lactating women and women of childbearing age do not take reliable contraceptive measures;
16. In the investigator's judgment, there is a concomitant medical condition (such as poorly controlled high blood pressure, severe diabetes, neurological or psychiatric illness, etc.) or any other condition that seriously endangers the subject's safety, may confuse the study results, or may interfere with the subject's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-16 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  ORR(objective response rate) is defined as the proportion of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator using RECIST 1.1.

SECONDARY OUTCOMES:
Progression Free Survival | 3 years
  PFS(progression-free survival), defined as the time from the date of randomization to the date of the first documentation of progressive disease (PD) or death (whichever occurred first)
Overall Survival | 3 years
  OS(overall survival) is defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No